CLINICAL TRIAL: NCT00539890
Title: A Phase 3 Randomized, Open Label, Multi-Center Comparative Study of Technosphere /Insulin Versus Rapid Acting Insulin in Subjects With Type-2 Diabetes Mellitus Receiving Lantus as Basal Insulin
Brief Title: Comparison Between Technosphere/Insulin Inhalation Powder Versus Rapid Acting Insulin in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-014
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Technosphere Insulin

SUMMARY:
To compare the efficacy of prandial TI plus basal insulin versus prandial rapid acting, subcutaneous insulin plus basal insulin in subjects with type 2 diabetes who had an HbA1c >7.0% and <11.5%.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 years since diagnosis of type 2 diabetes mellitus
* Received subcutaneous (sc) insulin for at least 3 months
* Body Mass Index <44 kg/m2
* HbA1c>7.0% and <11.5%
* Serum creatinine <2.0 mg/dL for males and <1.8 mg/dL for females
* Baseline FVC and FEV1>70% and < 125% of predicted normal

Exclusion Criteria:

* Significant hepatic disease (AST/ALT3 x ULN)
* Diagnosis of Type 1 diabetes
* Severe complications of diabetes
* History of moderate to severe ketoacidosis within the past 3 months
* Upper respiratory infection in the last 15 days or a lower respiratory infection in the past 30 days
* Diagnosis of HIV
* Positive serology for hepatitis B or C
* COPD, emphysema, or asthma
* Current smokers or smoking history within the past 6 months
* Major psychiatric disorder precluding satisfactory completion of protocol
* Clinically significant heart disease disease, stroke or heart attack within the past 6 months
* Treatment with an investigational drug within 30 days
* Previous treatment with Technosphere/Insulin
* History of malignancy in the past 5 years except basal cell carcinoma
* Anemia (hemoglobin <10.5 g/dL for females and <11.5 g/dL (for males)
* Women who were pregnant of lactating
* History of hypersensitivity to drugs resembling FDKP carrier products
* Treatment with another inhaled insulin product during the duration of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 2005-11; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c from baseline to treatment week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Baughman, PhD, Study Director — Mannkind Corporation
Locations (33):
- Russia (33):
  - Ural State Medical Academy of Post-Graduate Education Municipal Clinical Hospital # 3, Chelyabinsk, RUS
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - NI Principal Military Clinical Hospital n a academician N.N. Burdenko of the Ministry of Defense, Moscow, RUS
  - Moscow State Medico-Stomatological University City Hospital # 23, Moscow, RUS
  - Russian State Medical University, Moscow, RUS
  - Clinical Research Institute of Physic-Chemical Medicine Hospital # 29, Moscow, RUS
  - NEI HPE Moscow State University of Medicine and Dentistry of FAHSD City Clinical Hospital #70, Moscow, RUS
  - Russian State Medical University City Hospital # 4, Moscow, RUS
  - Russian Academy of Medical Sciences National Research Ctr for Endocrinology Institute of Diabetes, Moscow, RUS
  - Moscow Hospital of Glavmosstroy State Unitary Enterprise Medical Centre Medical Sanitary Unit #47, Moscow, RUS
  - Russian State Medical University Central Clinical Hospital Russian Science Academy, Moscow, RUS
  - Sechenov Moscow Medical Academy, Moscow, RUS
  - Moscow Medical Academy, Moscow, RUS
  - Moscow, RUS
  - SIH of Moscow City Clinical Hopsital #81 Endocrinology and Diabetology, Moscow, RUS
  - Moscow State Medical Stomatology University Municipal Hospital # 63 Endocrinology Diabetology, Moscow, RUS
  - Moscow City Clinical Hospital # 20, Moscow, RUS
  - Municipal Clinical Hospital #13, Moscow, RUS
  - Nizhni Novgorod regional hospital na Semashko, Nizhny Novgorod, RUS
  - St Petersburg NHI City Polytclinic #77 City Diabetological Center #4, Saint Petersburg, RUS
  - Central Medical Sanitary Unit #122, Saint Petersburg, RUS
  - SPb Diabetological Center, Saint Petersburg, RUS
  - St Petersburg NHI Municipal Multi-Speciality Hospital # 2, Saint Petersburg, RUS
  - St Petersburg Medical Academy St Elizabeth Hospital, Saint Petersburg, RUS
  - Pavlov State Medical Univ of St Petersburg, Saint Petersburg, RUS
  - City Outpatient Clinic # 34, Saint Petersburg, RUS
  - TUV Medico-Military Academy, Saint Petersburg, RUS
  - Center Diabetes LLC, Samara, RUS
  - Saratov City Outpatient Clinic # 20, Saratov, RUS
  - Saratov Medical University Faculty Therapy Chair Clinical Hospital # 3, Saratov, RUS
  - NEI HPE Smolensk State Medical Academy of FAHSD RNHI Smolensk Regional Clinical Hospital, Smolensk, RUS
  - MHI Clinical Hospital for Emergency Care na NV Soloviev, Yaroslavl, RUS
  - Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS